CLINICAL TRIAL: NCT05855018
Title: A Randomized, Open-label Phase I Clinical Study to Evaluate the Systemic Pharmacokinetics and Safety of Atropine Sulfate Eye Drops in Healthy Chinese Volunteers
Brief Title: A Study of Atropine Sulfate in Healthy Chinese Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhaoke (Hong Kong) Ophthalmology Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Organization: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZKO(HK)-ATP-202111
Record Dates: First submitted 2023-04-23; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atropine sulfate Concentration A (Experimental): Subjects will be treated with atropine sulfate eye drop (at dosage Concentration A), administered once daily (QD).
  Interventions: Drug: Atropine sulfate eye drops
- Atropine sulfate Concentration B (Experimental): Subjects will be treated with atropine sulfate eye drop (at dosage Concentration B), administered once daily (QD).
  Interventions: Drug: Atropine sulfate eye drops
- Atropine sulfate Concentration C (Experimental): Subjects will be treated with atropine sulfate eye drop (at dosage Concentration C), administered once daily (QD).
  Interventions: Drug: Atropine sulfate eye drops

INTERVENTIONS:
Drug: Atropine sulfate eye drops — One drop once daily
  Other Names: Atropine sulfate

SUMMARY:
To evaluate the systemic pharmacokinetics and the safety of atropine sulfate eye drops in healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized, open-label, phase I clinical study evaluating the systemic pharmacokinetics and safety of atropine sulfate eye drops in healthy Chinese volunteers.Three concentrations will be investigated, each concentration group must contain both male and female subjects, and each subject receives only one concentration of atropine sulfate eye drop in this study.

The three treatment arms are:

Atropine sulfate dose A (low concentration)

Atropine sulfate dose B (medium concentration)

Atropine sulfate dose C (high concentration)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject is a male or female Chinese with his/her biological parents and grandparents are of Chinese ethnicity, aged 18-45 (including cut-off value) at screening;
2. Subject with a body mass index (BMI) between 19.0-26.0kg/m2 (including cut-off value), male weight ≥50.0kg, female weight ≥45.0kg at screening and D0;
3. Subject is in good health, as determined by the investigator, based on medical history, no findings of clinical significant abnormalities at physical examination, vital signs, electrocardiogram and clinical laboratory tests at screening and D0;

Exclusion Criteria:

1. Subject with any eye with corrected visual acuity <1.0, clinically significant abnormal intraocular pressure, slit lamp and fundus examination.
2. Subject with history of eye diseases, including the history of internal eye surgery or laser surgery.
3. Subject with clinically significant history of the central nervous system, mental, cardiovascular, kidney, liver, respiratory, metabolic, and musculoskeletal system diseases etc., which may endanger the safety of the subject or affect the results of the study, as judged by the investigator.
4. Subject with clinically significant history of allergies, such as drug allergies, especially those who are allergic to any component of atropine sulfate eye drops.
5. On average, subject smokes more than 5 cigarettes per day or that who ex-smokes less than 3 months.
6. Subject has used any topical or systemic antimuscarinic/anticholinergic drugs (e.g., atropine, 1-hyoscyamine, tropicamide, chlorpheniramine, diphenhydramine, oxytropine, cyclic antidepressants, etc.) within 3 weeks before screening.
7. Subject has used any local or systemic drugs (including any prescription or over-the-counter drugs) within 2 weeks before screening.
8. Subject has participated in interventional clinical trials within 3 months before screening.
9. Subject who has worn contact lenses or cosmetic contact lenses within 1 weeks before screening.
10. Subject who is pregnant or breastfeeding.
11. The investigator believes that the subject is not suitable to participate in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | From 1 hour before administration to 24 hours after administration
  Measure the concentration of analyte in the blood to evaluate drug pharmacokinetics
Time of Cmax (Tmax) | From 1 hour before administration to 24 hours after administration
  Measure the concentration of analyte in the blood to evaluate drug pharmacokinetics
Time of half-life (t1/2) | From 1 hour before administration to 24 hours after administration
  Measure the concentration of analyte in the blood to evaluate drug pharmacokinetics
Area Under time-concentration Curve from 0 to last draw time (AUC0-t) | From 1 hour before administration to 24 hours after administration
  Measure the concentration of analyte in the blood to evaluate drug pharmacokinetics
Area Under time-concentration Curve from 0 to infinity time (AUC(0-∞)) | From 1 hour before administration to 24 hours after administration
  Measure the concentration of analyte in the blood to evaluate drug pharmacokinetics
Minimum concentration (Cmin) | From 1 hour before administration to 24 hours after administration
  Measure the concentration of analyte in the blood to evaluate drug pharmacokinetics
Volume of distribution (Vd) | From 1 hour before administration to 24 hours after administration
  Measure the concentration of analyte in the blood to evaluate drug pharmacokinetics
Elimination rate constant (Kel) | From 1 hour before administration to 24 hours after administration
  Measure the concentration of analyte in the blood to evaluate drug pharmacokinetics
Clearance (CL) | From 1 hour before administration to 24 hours after administration
  Measure the concentration of analyte in the blood to evaluate drug pharmacokinetics
Apparent Clearance (CL/F) | From 1 hour before administration to 24 hours after administration
  Measure the concentration of analyte in the blood to evaluate drug pharmacokinetics

SECONDARY OUTCOMES:
Slit-lamp eye examination results change from baseline to Day 7 | on Day 0 and Day 7
  Evaluate the anterior segment of the eye, including the eyelids, cornea, conjunctiva, anterior chamber, iris and lens, and record abnormalities
Fundoscopy eye examination results change from baseline to Day 7 | on Day 0 and Day 7
  Evaluate the condition of the fundus, including the vitreous body, optic disc, macula, peripheral retina and retinal blood vessels
Intraocular pressure change from baseline to Day 7 | on Day 0 and Day 7
  Use non-contact tonometer to measure intraocular pressure
Vision acuity change from baseline to Day 7 | on Day 0 and Day 7
  Using Best-corrected LogMAR scale
The mean change of pupil diameter from baseline to Day 7 | on Day 0 and Day 7
  Use ophthalmic biometry equipment to measure pupil diameter
The mean change of accommodation amplitude from baseline to Day 7 | on Day 0 and Day 7
  Use a Phoropter to measure the accommodation amplitude using the negative lens method

CONTACTS AND LOCATIONS:
Overall Officials: Christopher LEUNG, Principal Investigator — HKU Eye Centre
Locations (1):
- HKU Eye Centre, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No